CLINICAL TRIAL: NCT01660022
Title: A Phase I Study to Investigate the Safety, Tolerability & Pharmacokinetics of Co-administered Single Doses of OZ439 and Piperaquine to Healthy Subjects
Brief Title: Safety Tolerability & Pharmacokinetics of Co-administered Single Doses of OZ439 & Piperaquine to Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medicines for Malaria Venture (Other)
Collaborators: Cross Research S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: MMV_OZ439_12_002
Record Dates: First submitted 2012-08-06; First posted 2012-08-08 (Estimated); Results first posted 2015-01-21 (Estimated); Last update posted 2015-01-21 (Estimated); Status verified 2015-01

CONDITIONS: Healthy
Keywords: Healthy; Volunteers
MeSH Terms: interventions — piperaquine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (9):
- OZ439 100mg (Experimental): 100mg OZ439 single oral dose
  Interventions: Drug: 100mg OZ439 single oral dose
- OZ439 100 mg + PQP 160mg (Experimental): 100mg OZ439 single oral dose + 160mg Piperaquine single oral dose
  Interventions: Drug: 100mg OZ439 single oral dose; Drug: 160mg Piperaquine single oral dose
- OZ439 100 mg + PQP 480mg (Experimental): 100mg OZ439 single oral dose + 480mg Piperaquine single oral dose
  Interventions: Drug: 100mg OZ439 single oral dose; Drug: 480mg Piperaquine single oral dose
- OZ439 100 mg + PQP 1440mg (Experimental): 100mg OZ439 single oral dose + 1440mg Piperaquine single oral dose
  Interventions: Drug: 100mg OZ439 single oral dose; Drug: 1440mg Piperaquine single oral dose
- OZ439 300mg (Experimental): 300mg OZ439 single oral dose
  Interventions: Drug: 300 mg OZ439 single oral dose
- OZ439 300 mg + PQP 1440mg (Experimental): 300mg OZ439 single oral dose + 1440mg Piperaquine single oral dose
  Interventions: Drug: 300 mg OZ439 single oral dose; Drug: 1440mg Piperaquine single oral dose
- OZ439 800mg (Experimental): 800mg OZ439 single oral dose
  Interventions: Drug: 800 mg OZ439 single oral dose
- OZ439 800 mg + PQP 1440mg (Experimental): 800mg OZ439 single oral dose + 1440mg Piperaquine single oral dose
  Interventions: Drug: 1440mg Piperaquine single oral dose; Drug: 800 mg OZ439 single oral dose
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 100mg OZ439 single oral dose — 100mg OZ439 oral suspension single dose
  Other Names: OZ439
  Arms: OZ439 100 mg + PQP 1440mg; OZ439 100 mg + PQP 160mg; OZ439 100 mg + PQP 480mg; OZ439 100mg
Drug: Placebo — Placebo
  Arms: Placebo
Drug: 300 mg OZ439 single oral dose — 300mg OZ439 oral suspension single dose
  Other Names: OZ439
  Arms: OZ439 300 mg + PQP 1440mg; OZ439 300mg
Drug: 160mg Piperaquine single oral dose — 160 mg Piperaquine tablet
  Other Names: Piperaquine
  Arms: OZ439 100 mg + PQP 160mg
Drug: 480mg Piperaquine single oral dose — 480 mg Piperaquine tablet
  Other Names: Piperaquine
  Arms: OZ439 100 mg + PQP 480mg
Drug: 1440mg Piperaquine single oral dose — 1440 mg Piperaquine tablet
  Other Names: Piperaquine
  Arms: OZ439 100 mg + PQP 1440mg; OZ439 300 mg + PQP 1440mg; OZ439 800 mg + PQP 1440mg
Drug: 800 mg OZ439 single oral dose — 800mg OZ439 oral suspension single dose
  Other Names: OZ439
  Arms: OZ439 800 mg + PQP 1440mg; OZ439 800mg

SUMMARY:
A Phase I Study to investigate the safety, tolerability & pharmacokinetics of co-administered single doses of OZ439 and Piperaquine to healthy subjects.

DETAILED DESCRIPTION:
Placebo-controlled, double-blind, five-cohort, 2-period (per cohort) dose-escalation study.

For each subject, the study included a screening evaluation (within 21 days of the 1st dose), dosing on 2 separate occasions (Period 1 and Period 2) and a follow-up visit (6 weeks following the final dose).

Within each cohort, subjects were randomised into two sequences to receive OZ439 in Period 1 and OZ439 plus piperaquine in Period 2 (sequence 1, 8 subjects) or OZ439-matching placebo in Period 1 and OZ439/piperaquine matching placebos in Period 2 (sequence 2, 4 subjects).

Safety and tolerability were evaluated: Physical examination, ECG assessments including a full baseline matched profile of ECG tracings, vital signs, laboratory evaluations, in particular liver function tests and adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males & females, 18-55 years old
* BMI 18 to 30kg/m2; total body weight >50kg
* Healthy, determined by pre-study medical history, physical examination vital signs, 12 Lead ECG
* Females of non-childbearing potential.
* Males must agree to use a double barrier method of contraception
* Lab tests at screening within the reference ranges

Exclusion Criteria:

* Any condition that could affect drug absorption, e.g. gastrectomy, diarrhea
* Clinically relevant abnormalities in ECG
* Family history of sudden death or of congenital prolongation of QTc interval - History of symptomatic cardiac arrhythmias or with clinically relevant bradycardia
* Electrolyte disturbances
* History of drug or alcohol abuse, tobacco users
* Participation in evaluation of any drug for 3 months before the study
* Administration of ANY systemic medication/herbal product within 14 days of first dose of study drug.
* unaccustomed strenuous exercise within 7 days of any study visit
* Alcohol consumption within 24 hours of any study visit
* Consumption of any fruit juice or food containing grapefruit within 7 days
* Positive test for HIV-1, HBsAg or HCV
* Positive urine drug screen at Screening or admission
* Severe allergies/multiple drug allergies
* Volunteers who have donated blood or experienced significant blood loss within 90 days of screening
* Hemoglobin below lower limit of the reference range
* Clinically relevant abnormal lab values indicative of physical illness

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2012-09; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Milko M Radicioni, MD PhD, Principal Investigator — Cross Research S.A.
Locations (1):
- Cross Research S.A., Mendrisio, Switzerland

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Date of first enrolment: 11SEP2012 Date last volunteer completed: 07MAY2013 Phase 1 Clinical Research Unit
Groups:
- Cohort 1: Sequence 1: OZ439 100mg Sequence 2: OZ439 100mg / PQP 160mg
- Cohort 2: Sequence 1: OZ439 100mg Sequence 2: OZ439 100mg+PQP 480mg
- Cohort 3: Sequence 1: OZ439 100mg Sequence 2: OZ439 100mg+PQP 1440mg
- Cohort 4: Sequence 1: OZ439 300mg Sequence 2: OZ439 300mg+PQP 1440mg
- Cohort 5: Sequence 1: OZ439 800mg Sequence 2: OZ439 800mg+PQP 1440mg
- Placebo: Cohorts 1, 2, 3, 4 and 5
Period: First Sequence (7 Days)
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Placebo
Started | 8 | 8 | 8 | 8 | 7 | 20
Completed | 8 | 7 | 8 | 7 | 6 | 16
Not Completed | 0 | 1 | 0 | 1 | 1 | 4
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 3
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 1
Period: Second Sequence (42 Days)
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Placebo
Started | 8 | 7 | 8 | 7 | 6 | 16
Completed | 8 | 7 | 8 | 7 | 6 | 16
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population
Groups:
- Cohort 1: Sequence 1: OZ439 100mg Sequence 2: OZ439 100 mg / PQP 160 mg
- Cohort 2: Sequence 1: OZ439 100mg Sequence 2: OZ439 100 mg / PQP 480 mg
- Cohort 3: Sequence 1: OZ439 100mg Sequence 2: OZ439 100 mg / PQP 1440 mg
- Cohort 4: Sequence 1: OZ439 300mg Sequence 2: OZ439 300 mg / PQP 1440 mg
- Cohort 5: Sequence 1: OZ439 800mg Sequence 2: OZ439 800 mg / PQP 1440 mg
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Placebo | Total
Number analyzed (Participants) | 8 | 7 | 8 | 7 | 6 | 20 | 56
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.0 (9.4) | 41.7 (7.1) | 35.4 (10) | 32.1 (8.4) | 35.7 (11.7) | 37.3 (10.3) | 36.43 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Male | 8 | 7 | 8 | 7 | 6 | 19 | 55
Region of Enrollment [Number; unit: participants]
  Switzerland | 8 | 7 | 8 | 7 | 6 | 20 | 56

OUTCOME MEASURES:

1. Primary Outcome: OZ439 Cmax
Description: OZ439 Maximum concentration level
Time Frame: Up to 168 hours post-dose
Population: All randomised subjects who fulfilled the study protocol requirements in terms of study drug intake and PK samplings, with no major deviations that could affect the PK results.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Cohort 1 - OZ439 100mg: Cohort 1 - Sequence 1 OZ439 100mg
- Cohort 1 - OZ439 100mg / PQP 160mg: Cohort 1 - Sequence 2 OZ439 100mg / PQP 160mg
- Cohort 2 - OZ439 100mg: Cohort 2 - Sequence 1 OZ439 100mg
- Cohort 2 - OZ439 100mg / PQP 480mg: Cohort 2 - Sequence 2 OZ439 100mg / PQP 480mg
- Cohort 3 - OZ439 100mg: Cohort 3 - Sequence 1 OZ439 100mg
- Cohort 3 - OZ439 100mg / PQP 1440mg: Cohort 3 - Sequence 2 OZ439 100mg / PQP 1440mg
- Cohort 4 - OZ439 300mg: Cohort 4 - Sequence 1 OZ439 300mg
- Cohort 4 - OZ439 300mg / PQP 1440mg: Cohort 4 - Sequence 2 OZ439 300mg / PQP 1440mg
- Cohort 5 - OZ439 800mg: Cohort 5 - Sequence 1 OZ439 800mg
- Cohort 5 - OZ439 800mg / PQP 1440mg: Cohort 5 - Sequence 2 OZ439 800mg / PQP 1440mg
Arm/Group | Cohort 1 - OZ439 100mg | Cohort 1 - OZ439 100mg / PQP 160mg | Cohort 2 - OZ439 100mg | Cohort 2 - OZ439 100mg / PQP 480mg | Cohort 3 - OZ439 100mg | Cohort 3 - OZ439 100mg / PQP 1440mg | Cohort 4 - OZ439 300mg | Cohort 4 - OZ439 300mg / PQP 1440mg | Cohort 5 - OZ439 800mg | Cohort 5 - OZ439 800mg / PQP 1440mg
Number analyzed (Participants) | 8 | 8 | 7 | 7 | 8 | 8 | 7 | 7 | 5 | 5
ng/mL | 142 (39.2) | 139 (33.1) | 146 (43.2) | 198 (47.4) | 127 (22.9) | 199 (26.8) | 590 (31.5) | 778 (31.5) | 1500 (42.2) | 1650 (25.6)

2. Primary Outcome: Piperaquine Cmax
Description: Piperaquine Maximum concentration level
Time Frame: Up to 1008 hours post-dose (Day 43)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- OZ439 100mg / PQP 160mg: Cohort 1 - Sequence 2 OZ439 100mg / PQP 160mg
- OZ439 100mg / PQP 480mg: Cohort 2 - Sequence 2 OZ439 100mg / PQP 480mg
- OZ439 100mg / PQP 1440mg: Cohort 3 - Sequence 2 OZ439 100mg / PQP 1440mg
- OZ439 300mg / PQP 1440mg: Cohort 4 - Sequence 2 OZ439 300mg / PQP 1440mg
- OZ439 800mg / PQP 1440mg: Cohort 5 - Sequence 2 OZ439 800mg / PQP 1440mg
Arm/Group | OZ439 100mg / PQP 160mg | OZ439 100mg / PQP 480mg | OZ439 100mg / PQP 1440mg | OZ439 300mg / PQP 1440mg | OZ439 800mg / PQP 1440mg
Number analyzed (Participants) | 8 | 7 | 8 | 7 | 5
ng/mL | 8.59 (34.7) | 46.6 (44.3) | 393 (43.8) | 271 (30.9) | 356 (53.6)

3. Primary Outcome: OZ439 AUC(0-168)
Description: Area under the plasma concentration versus time curve to 168 hours post-dose.
Time Frame: Up to 168 hours post-dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng.h/mL
Arm/Group | Cohort 1 - OZ439 100mg | Cohort 1 - OZ439 100mg / PQP 160mg | Cohort 2 - OZ439 100mg | Cohort 2 - OZ439 100mg / PQP 480mg | Cohort 3 - OZ439 100mg | Cohort 3 - OZ439 100mg / PQP 1440mg | Cohort 4 - OZ439 300mg | Cohort 4 - OZ439 300mg / PQP 1440mg | Cohort 5 - OZ439 800mg | Cohort 5 - OZ439 800mg / PQP 1440mg
Number analyzed (Participants) | 8 | 8 | 7 | 7 | 8 | 8 | 7 | 7 | 5 | 5
ng.h/mL | 862 (33.9) | 920 (26.6) | 1130 (41.7) | 1390 (47.0) | 909 (21.4) | 1520 (26.1) | 5740 (29.9) | 7410 (30.3) | 15300 (47.6) | 18600 (36.8)

4. Primary Outcome: OZ439 t1/2
Description: OZ439 Elimination half-life
Time Frame: Up to 168 hours post-dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour
Arm/Group | Cohort 1 - OZ439 100mg | Cohort 1 - OZ439 100mg / PQP 160mg | Cohort 2 - OZ439 100mg | Cohort 2 - OZ439 100mg / PQP 480mg | Cohort 3 - OZ439 100mg | Cohort 3 - OZ439 100mg / PQP 1440mg | Cohort 4 - OZ439 300mg | Cohort 4 - OZ439 300mg / PQP 1440mg | Cohort 5 - OZ439 800mg | Cohort 5 - OZ439 800mg / PQP 1440mg
Number analyzed (Participants) | 8 | 8 | 7 | 7 | 8 | 8 | 7 | 7 | 5 | 5
hour | NA (NA) — Insufficient data points for calculation | NA (NA) — Insufficient data points for calculation | NA (NA) — Insufficient data points for calculation | NA (NA) — Insufficient data points for calculation | NA (NA) — Insufficient data points for calculation | NA (NA) — Insufficient data points for calculation | 90.6 (19.4) | 112 (45.2) | 65.4 (23.2) | 135 (53.2)

5. Primary Outcome: Piperaquine AUC(0-168)
Description: Piperaquine area under the plasma concentration versus time curve to 168 hours post-dose
Time Frame: Up to 1008 hours post-dose (Day 43)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng.h/mL
Arm/Group | OZ439 100mg / PQP 160mg | OZ439 100mg / PQP 480mg | OZ439 100mg / PQP 1440mg | OZ439 300mg / PQP 1440mg | OZ439 800mg / PQP 1440mg
Number analyzed (Participants) | 8 | 7 | 8 | 7 | 5
ng.h/mL | 1340 (NA) — Not Calculated. Insufficient data points for calculation. | 3420 (22.8) | 17500 (25.7) | 17200 (12.8) | 13200 (53.8)

6. Primary Outcome: Piperaquine t1/2
Description: Piperaquine Elimination half-life (t1/2).
Time Frame: Up to 1008 hours post-dose (Day 43)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour
Arm/Group | OZ439 100mg / PQP 160mg | OZ439 100mg / PQP 480mg | OZ439 100mg / PQP 1440mg | OZ439 300mg / PQP 1440mg | OZ439 800mg / PQP 1440mg
Number analyzed (Participants) | 8 | 7 | 8 | 7 | 5
hour | 294 (NA) — Not Calculated. Insufficient data points for calculation. | 283 (64.4) | 515 (36.3) | 632 (26.5) | 509 (15.9)

ADVERSE EVENTS:
Time Frame: From informed consent signature up to final study visit.
Description: Safety variables: treatment-emergent adverse events (TEAEs), ECG results, vital signs, laboratory evaluations, in particular liver function tests.
Groups:
- OZ439 100mg: Cohorts 1, 2 and 3 OZ439 100mg
- OZ439 300mg: Cohort 4 - Sequence 1 OZ439 300mg
- OZ439 800mg: Cohort 5 - Sequence 1 OZ439 800mg
Arm/Group | OZ439 100mg | OZ439 300mg | OZ439 800mg | OZ439 100mg / PQP 160mg | OZ439 100mg / PQP 480mg | OZ439 100mg / PQP 1440mg | OZ439 300mg / PQP 1440mg | OZ439 800mg / PQP 1440mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/8 | 0/7 | 0/8 | 0/7 | 0/8 | 0/7 | 0/6 | 1/20
Other Adverse Events (participants affected / at risk) | 3/24 | 3/8 | 2/7 | 2/8 | 0/7 | 1/8 | 3/7 | 1/6 | 8/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OZ439 100mg (N=24) | OZ439 300mg (N=8) | OZ439 800mg (N=7) | OZ439 100mg / PQP 160mg (N=8) | OZ439 100mg / PQP 480mg (N=7) | OZ439 100mg / PQP 1440mg (N=8) | OZ439 300mg / PQP 1440mg (N=7) | OZ439 800mg / PQP 1440mg (N=6) | Placebo (N=20)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Eosinophilia (55% ; 9.81 g/l). Concomitant medication taken; hospitalization/prolonged hospitalization. Outcome: Recovery
OTHER ADVERSE EVENTS (reported when occurring in more than 4.17% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OZ439 100mg (N=24) | OZ439 300mg (N=8) | OZ439 800mg (N=7) | OZ439 100mg / PQP 160mg (N=8) | OZ439 100mg / PQP 480mg (N=7) | OZ439 100mg / PQP 1440mg (N=8) | OZ439 300mg / PQP 1440mg (N=7) | OZ439 800mg / PQP 1440mg (N=6) | Placebo (N=20)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) — Eosinophilia
Abdominal Discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) — Abdominal Discomfort
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Diarrhea
Gastroenteritis Eosinophilic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Gastroenteritis Eosinophilic
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) — Nausea
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) — Vomiting
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Malaise
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) — Nasopharyngitis Pathogen Unspecified
ALT Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) — ALT Increased
AST Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — AST Increased
Blood Creatine Phosphokinase increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (5) — Blood Creatine Phosphokinase increased
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Hypercalcaemia
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Hyperkalaemia
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Back Pain
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Headache

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days